CLINICAL TRIAL: NCT03733405
Title: Randomized Control Trial of Postpartum Visits at Two or Six Weeks to Evaluate Clinic Attendance and Emergency Department Usage
Brief Title: Postpartum Care Timing: A Randomized Trial
Acronym: PUnCTuAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Ilina Datkhaeva, Co-principal investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18-001453
Record Dates: First submitted 2018-11-05; First posted 2018-11-07 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Postpartum; Pregnancy Related
Keywords: Breastfeeding; Contraception; Emergency; Department
MeSH Terms: conditions — Breast Feeding; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postpartum Visit 6 Weeks (Experimental): Participants will have a postpartum visit scheduled 6 weeks after birth
  Interventions: Behavioral: Postpartum Visit at 6 Weeks
- Postpartum Visit 2 and 6 Weeks (Experimental): Participants will have postpartum visits scheduled 2 and 6 weeks after birth
  Interventions: Behavioral: Postpartum Visit at 6 Weeks; Behavioral: Postpartum Visit at 2 Weeks

INTERVENTIONS:
Behavioral: Postpartum Visit at 6 Weeks — The patient will be scheduled for a routine postpartum visit at the standard time interval. Each postpartum visit will consist of the standard interview and physical examination. The purpose of this visit is for routine postpartum care. If she has a medical complication during delivery, she may be recommended to schedule an additional earlier visit.
Behavioral: Postpartum Visit at 2 Weeks — The patient will be scheduled for an earlier postpartum visit in addition to the standard time interval. Each postpartum visit will consist of the standard interview and physical examination. The purpose of this visit is for routine postpartum care. If she has a medical complication during delivery, she may be recommended to schedule an additional earlier visit.
  Arms: Postpartum Visit 2 and 6 Weeks

SUMMARY:
The purpose of this study is to determine if shortening the time to initial postpartum visit from six weeks to two weeks can improve clinic visit attendance and decrease usage of the emergency department.

DETAILED DESCRIPTION:
Postpartum care is an integral component to completing the maternal peripartum experience and transitioning the patient to well-women care. The American Congress of Obstetrics and Gynecology has recently highlighted the importance of this "fourth stage" of pregnancy suggesting earlier and more comprehensive visits compared to the standard 6-week postpartum visit. Specifically they describe that "all women should ideally have contact with a maternal care provider within the first three weeks postpartum" however this is largely derived from expect opinion and retrospective data. The current rate of postpartum visit attendance is as low as 66%, especially in women with scant prenatal care. In the investigators government-funded clinic, the postpartum clinic attendance in 2017 was 69% and many of the patients have co-morbidities, notably a 25% rate of psychiatric illness. Additionally, in this population, the investigators have identified a high rate of Emergency Department (ED) usage (8.7%) within 30 days of delivery suggesting that perhaps an earlier routine visit is ideal and can prevent the use of the ED. The aim therefore is to evaluate the utility of an early postpartum visit at two weeks in addition to a standard six-week visit with a randomized control trial.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Receives antepartum, intrapartum and postpartum care at UCLA
* Speaks English or Spanish
* Provides informed consent for study participation
* Vaginal, cesarean delivery or operative vaginal delivery

Exclusion Criteria:

* Cognitive impairment, psychiatric instability, or language barriers that limit her ability to provide informed consent
* Plans to received postpartum care at other institution

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 256 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Attendance at one or more routine postpartum visits | 8 weeks postpartum
  The primary outcome will be the attendance at one or more scheduled postpartum visits at the clinic where the patient received her prenatal care.

SECONDARY OUTCOMES:
Rate of Emergency Department usage within 30 days of delivery | 30 days postpartum
  The secondary outcome will be the presentation and usage of an Emergency Department during the 30 days since delivery of the baby.

CONTACTS AND LOCATIONS:
Overall Officials: Ilina Datkhaeva, MD, Study Director — University of California, Los Angeles
Locations (1):
- University of California Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pluym ID, Tandel MD, Kwan L, Mok T, Holliman K, Afshar Y, Rao R. Randomized control trial of postpartum visits at 2 and 6 weeks. Am J Obstet Gynecol MFM. 2021 Jul;3(4):100363. doi: 10.1016/j.ajogmf.2021.100363. Epub 2021 Mar 27. PMID 33785465